CLINICAL TRIAL: NCT05361395
Title: A Phase 1b Study Evaluating the Safety and Efficacy of First-Line Tarlatamab in Combination With Carboplatin, Etoposide, and PD-L1 Inhibitor in Subjects With Extensive Stage Small Cell Lung (DeLLphi-303)
Brief Title: First-Line Tarlatamab in Combination With Carboplatin, Etoposide, and PD-L1 Inhibitor in Subjects With Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200469; 2024-511021-58 (EudraCT Number)
Expanded Access: NCT06064500 (Approved for marketing)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Extensive Stage Small Cell Lung Cancer; ES-SCLC; SCLC; Lung Cancer; AMG 757; Bi-Specific T-Cell Engager; BiTE; Inmunotherapy; Immunooncology; Inmuno-oncology; DLL3; Delta Like Protein 3
MeSH Terms: conditions — Lung Neoplasms; Bites and Stings | interventions — AMG 757; Carboplatin; Etoposide; atezolizumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Dose Exploration Combination Regimen 1 (Experimental): Tarlatamab+Atezolizumab+Carboplatin+Etoposide
  Interventions: Drug: Tarlatamab; Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab
- Part 2: Dose Exploration Combination Regimen 2 (Experimental): Tarlatamab+Atezolizumab+Carboplatin+Etoposide
  Interventions: Drug: Tarlatamab; Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab
- Part 3: Dose Exploration Combination Regimen 3 (Experimental): Tarlatamab+Atezolizumab+Carboplatin+Etoposide
  Interventions: Drug: Tarlatamab; Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab
- Part 4: Dose Expansion (Experimental): Expansion of Part 1, Part 2, or Part 3 with Atezolizumab
  Interventions: Drug: Tarlatamab; Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab
- Part 5: Dose Exploration Maintenance (Experimental): Tarlatamab+Atezolizumab
  Interventions: Drug: Tarlatamab; Drug: Atezolizumab
- Part 6: Dose Expansion Maintenance (Experimental): Expansion of Part 5 with Atezolizumab
  Interventions: Drug: Tarlatamab; Drug: Atezolizumab
- Part 7: Dose Expansion (Experimental): Expansion of Part 1, 2, or 3 with Durvalumab
  Interventions: Drug: Tarlatamab; Drug: Carboplatin; Drug: Etoposide; Drug: Durvalumab
- Part 8: Dose Expansion Maintenance (Experimental): Expansion of Part 5 with Durvalumab
  Interventions: Drug: Tarlatamab; Drug: Durvalumab
- Part 9: Dose Expansion Maintenance (Experimental): Expansion with Tarlatamab+Durvalumab
  Interventions: Drug: Tarlatamab; Drug: Durvalumab

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered as an intravenous (IV) infusion.
  Other Names: AMG 757
Drug: Carboplatin — Carboplatin will be administered as an intravenous (IV) infusion.
  Arms: Part 1: Dose Exploration Combination Regimen 1; Part 2: Dose Exploration Combination Regimen 2; Part 3: Dose Exploration Combination Regimen 3; Part 4: Dose Expansion; Part 7: Dose Expansion
Drug: Etoposide — Etoposide will be administered as an intravenous (IV) infusion.
  Arms: Part 1: Dose Exploration Combination Regimen 1; Part 2: Dose Exploration Combination Regimen 2; Part 3: Dose Exploration Combination Regimen 3; Part 4: Dose Expansion; Part 7: Dose Expansion
Drug: Atezolizumab — Atezolizumab will be administered as an intravenous (IV) infusion.
  Other Names: Tecentriq
  Arms: Part 1: Dose Exploration Combination Regimen 1; Part 2: Dose Exploration Combination Regimen 2; Part 3: Dose Exploration Combination Regimen 3; Part 4: Dose Expansion; Part 5: Dose Exploration Maintenance; Part 6: Dose Expansion Maintenance
Drug: Durvalumab — Durvalumab will be administered as an intravenous (IV) infusion.
  Arms: Part 7: Dose Expansion; Part 8: Dose Expansion Maintenance; Part 9: Dose Expansion Maintenance

SUMMARY:
This is a phase 1b study to assess the safety and tolerability of tarlatamab in combination with programmed death ligand (PD-L1) inhibition with and without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age greater than or equal to 18 years old at the same time of signing the informed consent.
* Histologically or cytologically confirmed Extensive Stage Small Cell Lung Cancer (ES-SCLC) and no prior systemic treatment for ES-SCLC.
* Participants with prior treatment for limited-stage SCLC (LS-SCLC) are permitted.
* Eastern Cooperative Oncology Group (ECOG) 0 to 1.
* Participants with treated asymptomatic brain metastases are eligible provided they meet defined criteria.
* Adequate organ function as defined in protocol.

Exclusion Criteria:

* History of other malignancy within the past 2 years with exceptions.
* Major surgery within 28 days of study day 1.
* Untreated or symptomatic brain metastases and leptomeningeal disease.
* Participants who experienced recurrent grade 2 pneumonitis or severe or life-threatening immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents.
* History of immune-related colitis.
* History or evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Participants with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment
* Participant has known active infection requiring parenteral antibiotic treatment. Upon completion of parenteral antibiotics and resolution of symptoms, the participant may be considered eligible for the study from an infection standpoint
* NOTE: Simple urinary tract infections and uncomplicated bacterial pharyngitis are permitted if responding to an active treatment and after consultation with Medical Monitor. Participants requiring oral antibiotics who have been afebrile for >24 hours, have no leukocytosis, nor clinical signs of infection are eligible. Screening for chronic infectious conditions is not required.
* History of hypophysitis or pituitary dysfunction.
* History of solid organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study. Participants with Type I diabetes, vitiligo, psoriasis, hypo- or hyper-thyroid disease not requiring immunosuppressive treatment are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2028-08-28 (Estimated); Study Completion 2028-08-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Dose Limiting Toxicity (DLT) | 24 months
Number of Participants with Treatment-emergent Adverse Events (TEAE) | 24 months
Number of Participants with Treatment-related Adverse Events | 24 months
Number of Participants with Clinically Significant Changes in Vital Signs | 24 months
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Measurements | 24 months
Number of Participants with Clinically Significant Changes in Clinical Laboratory Tests | 24 months

SECONDARY OUTCOMES:
6-month Progression-free Survival (PFS) | 24 months
Objective Response (OR) | 24 months
  Per modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Duration of Response (DOR) | 24 months
Disease Control Rate(DCR) | 24 months
Overall Survival (OS) | 24 months
Serum Concentration of Tarlatamab | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (44):
- United States (9):
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Christiana Care Health Services, Newark, Delaware
  - Henry Ford Health System, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Grossman School of Medicine and New York University Langone Hospitals, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Swedish Cancer Institute Medical Oncology, Seattle, Washington
  - West Virginia University Health Sciences Center, Morgantown, West Virginia
- Chris OBrien Lifehouse, Camperdown, New South Wales, Australia
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - AZ Delta Campus Rumbeke, Roeselare
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Quebec Hopital de l Enfant Jesus, Québec, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire de Nantes, Hôpital Nord Laënnec, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (3):
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro
  - Fondazione IRCCS San Gerardo dei Tintori, Monza (MB)
  - Istituto Nazionale Tumori Regina Elena, Rome
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Institut Catala d Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (2):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Paulson KG, Lau SCM, Ahn MJ, Moskovitz M, Pogorzelski M, Hafliger S, Parkes A, Zhang Y, Hamidi A, Thompson CG, Wermke M. Safety and activity of tarlatamab in combination with a PD-L1 inhibitor as first-line maintenance therapy after chemo-immunotherapy in patients with extensive-stage small-cell lung cancer (DeLLphi-303): a multicentre, non-randomised, phase 1b study. Lancet Oncol. 2025 Oct;26(10):1300-1311. doi: 10.1016/S1470-2045(25)00480-2. Epub 2025 Sep 8. PMID 40934933
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com